CLINICAL TRIAL: NCT05171387
Title: A Single-arm, Open-label Phase 2 Study of Darolutamide in Addition to Standard Androgen Deprivation Therapy (ADT) in Chinese Participants With High-risk Non-metastatic Castration-resistant Prostate Cancer (nmCRPC)
Brief Title: Darolutamide + Androgen Deprivation Therapy (ADT) in Chinese Men With High Risk, Nonmetastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20963
Record Dates: First submitted 2021-10-22; First posted 2021-12-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Non-metastatic; castration resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Treatment period: The start of the treatment period is defined by the first administration of the study treatment (Day 1). The participants will take 2 tablets (300 mg each tablet) of study treatment (darolutamide) orally BID at about 12- hour intervals. All participants must also continue ADT treatment if they have not had bilateral orchiectomy. Doses of study treatment may be modified in case of clinically significant toxicities. Participants will receive study treatment until any of the discontinuation criteria are met.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Darolutamide in addition to Androgen deprivation therapy (Experimental)
  Interventions: Drug: Darolutamide 600 mg twice daily; Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Darolutamide 600 mg twice daily — The participants will take 2 tablets (300 mg each tablet) of study treatment (darolutamide) orally bid at about 12 hour intervals.
Drug: Androgen deprivation therapy (ADT) — Androgen deprivation therapy (ADT) is a treatment that commonly used to lower the amount of hormones called androgens in the body.

SUMMARY:
Researchers are seeking better ways to treat men who have non-metastatic castration resistant prostate cancer (nmCRPC). This type of prostate cancer-nmCRPC- is one that has not spread to other parts of the body yet keeps progressing despite low levels of (the hormone) testosterone. Signs of cancer progression are detected by higher (blood) levels of a protein known as "prostate-specific antigen" (PSA). PSA is made by both normal and cancerous cells in the body. An established treatment that is used to lower the amount of androgen hormones (e.g., testosterone) in the body is known as "Androgen deprivation therapy" (ADT), and all study participants will receive this (if they have not had surgery to remove their testicles). All participants will also receive the study-drug, darolutamide, which is already available for doctors to prescribe to patients with this condition. Darolutamide works by blocking the attachment of androgen hormones to androgen receptors in cancer cells, thereby blocking cancer progression and growth. There has been a previous research study that showed that patients with nmCRPC benefit from the combination of darolutamide plus Androgen deprivation therapy (ADT) when compared with placebo plus ADT therapy. Participants from mainland China were not included in the previous study.

The present study focuses specifically on Chinese participants with nmCRPC, who will receive both medications- darolutamide plus ADT. Researchers will be using a "marker" of cancer- PSA- to look at how the PSA declines when participants take study treatment. By using the tumor marker PSA, researchers can more quickly identify how study participants are responding to their study treatment. All the participants will also take ADT.

During the study, participants will take darolutamide until: (1) their cancer spreads (2) they start another type of cancer treatment (3) they have an adverse event that requires stopping the medication. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events is related to the study treatments. Other reasons for study discontinuation include: (4) a participant takes another type of medication that is not permitted to be taken during this study (5) the patient chooses to leave the trial or (6) the participant dies.

Study participants will visit the study site every 12 weeks for the first 3 visits and after visit 3, visit interval will be every 16 weeks during treatment and after stopping treatment (participants may continue to be followed even after stopping treatment). It is anticipated that the whole study will last about 35 months. During the study, doctors will: (1) check the participants' overall health and heart health (2) take blood samples (3) take pictures of the participants' tumors and bones using CT, MRI, and bone scans and (4) ask the participants questions about how they are feeling, what medications they are taking, and about adverse events they might be having.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age inclusive, at the time of signing the informed consent.
* Histologically or cytologically confirmed adenocarcinoma of prostate without neuroendocrine differentiation or small cell features.
* Castration resistance, demonstrated by:

  * a minimum of 3 rising PSA values while the participant is on continuous ADT (started at least 4 weeks prior to the PSA measurement or, PSA measured at least 4 weeks after bilateral orchiectomy) and
  * the interval between each PSA measurement must be ≥1 week, and
  * the PSA value at screening must be ≥1 ng/mL (1 μg/L). (To confirm this eligibility criterion, it is acceptable for 2 out of the 3 PSA measurements to be taken during the 28-day screening period (after participant has signed consent), provided the measurements are ≥1 week apart. In this case, the last PSA value should be recorded as the screening value.)
* Castrate level of serum testosterone (< 1.7 nmol/l [50 ng/dl]) on GnRH agonist or antagonist therapy or after bilateral orchiectomy. Participants who have not undergone bilateral orchiectomy must continue GnRH therapy during the study.
* Prostate-specific antigen doubling time (PSADT) of ≤ 10 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Blood counts at screening: hemoglobin ≥ 9.0 g/dl, absolute neutrophil count ≥ 1500/μl (1.5x109/l), platelet count ≥ 100,000/μl (100x109/l ) (participant must not have received any growth factor or blood transfusion within 7 days of the hematology laboratory obtained at screening).
* Screening values of serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN), total bilirubin (TBL) ≤1.5 x ULN (except participants with a diagnosis of Gilbert's disease), creatinine ≤2.0 x ULN.
* Male: Sexually active participants, unless surgically sterile, must agree to use condoms as an effective barrier method and refrain from sperm donation during the study treatment and for 1 week after the end of the study treatment. If the participant is engaged in sexual activity with a woman of childbearing potential (WOCBP), highly effective contraception should be used during and for 1 week after completion of treatment with darolutamide to prevent pregnancy.Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* History of metastatic disease at any time or presence of detectable metastases assessed by the investigator within 42 days prior to start of study treatment. Presence of pelvic lymph nodes < 1.5 cm in short axis below the aortic bifurcation is allowed.
* Symptomatic local-regional disease that requires medical intervention including moderate/severe urinary obstruction or hydronephrosis due to prostate cancer.
* Acute toxicities of prior treatments and procedures not resolved to ≤ CTCAE v5.0 grade 1 or baseline before treatment assignment.
* Severe or uncontrolled concurrent disease, infection or co-morbidity that, in the opinion of the investigator, would make the participant inappropriate for enrollment.
* Known hypersensitivity to the study treatment or any of its ingredients.
* Major surgery within 28 days before treatment assignment.
* Any of the following within 6 months before treatment assignment: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV.
* Uncontrolled hypertension as indicated by a systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite medical management at screening.
* Prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e. pTis, pTa, and pT1) is allowed, as well as any other cancer for which treatment has been completed ≥ 5 years ago and from which the participant has been disease-free.
* Gastrointestinal disorder or procedure which expects to interfere significantly with absorption of study treatment.
* Active viral hepatitis, known human immunodeficiency virus (HIV) infection with detectable viral load, or chronic liver disease with a need of treatment.
* Any condition that in the opinion of the investigator would impair the participants' ability to comply with the study procedures.
* Unable to swallow study medications and/or comply with study requirements.
* Prior treatment with:

  * second-generation AR inhibitors such as enzalutamide, apalutamide, darolutamide, other investigational AR inhibitors
  * CYP17 enzyme inhibitor such as abiraterone acetate, TAK-700
  * Oral ketoconazole longer than for 28 days (continuous use).
* Use of estrogens or 5-α reductase inhibitors (finasteride, dutasteride) within 28 days before start of study treatment (Day 1) or first-generation AR inhibitors (bicalutamide, flutamide, nilutamide, cyproterone acetate) within 28 days before start of study treatment (Day 1).
* Prior chemotherapy or immunotherapy for prostate cancer, except adjuvant/neoadjuvant treatment completed > 2 years before teatment assignment.
* Use of systemic corticosteroid with dose greater than the equivalent 10 mg of prednisone/day within 28 days before start of treatment assignment.
* Radiation therapy (external beam radiation therapy [EBRT], brachytherapy, or radiopharmaceuticals) within 12 weeks before randomization.
* Treatment with an osteoclast-targeted therapy (bisphosphonate or denosumab) to prevent skeletal-related events within 12 weeks before randomization. Participants receiving osteoclast-targeted therapy to prevent bone loss at a dose and schedule indicated for osteoporosis may continue treatment at the same dose and schedule.
* Treatment with any investigational drug within 28 days before start of study treament (Day 1).
* Treatment with any investigational drug, or Traditional Chinese Medication (TCM) that is approved as a cancer treatment, within 28 days before start of study treatment (Day 1).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) response rate of ≥50% decline (PSA50) | The baseline PSA value will be the latest measurement prior to start of study treatment. A PSA decline of ≥50% must be confirmed by a second value obtained at least 3 weeks later
  PSA response rate of ≥50% decline is defined as the proportion of participants who have achieved a decline of 50% or more from baseline during treatment at any time.

SECONDARY OUTCOMES:
Number of participants with: Adverse events (AEs) and serious adverse events (SAEs) | Up to 30 days after the last dose of treatment
Number of participants with: Discontinuations and dose modifications of study treatment due to AEs | Up to 30 days after the last dose of treatment
Number of participants with: Laboratory abnormalities reported as AEs | Up to 30 days after the last dose of treatment
  The investigator must review the laboratory report, document this review, and record any changes that are clinically relevant based on his/her clinical judgement, occurring during the study in the AE section of the CRF.
Number of participants with: Changes in Electrocardiograms (ECGs) reported as AEs | Up to 30 days after the last dose of treatment
Number of participants with: Changes in physical examination outcomes reported as AEs | Up to 30 days after the last dose of treatment
Number of participants with: Changes in Eastern Cooperative Oncology Group (ECOG) performance status | Up to 30 days after the last dose of treatment
PSA response rate of ≥90% decline (PSA90) | A PSA decline of ≥90% must be confirmed by a second value obtained at least 3 weeks later.
  PSA response rate of ≥90% decline is defined as the proportion of participants who have achieved a decline of 90% or more from baseline during treatment at any time.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.